CLINICAL TRIAL: NCT02564341
Title: Collaborative Care Intervention to Improve Providers' Opioid Prescribing for HIV-infected Patients - Intervention Component
Brief Title: Targeting Effective Analgesia in Clinics for HIV - Intervention
Acronym: TEACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Emory University (Other); Grady Health System (Other)
Responsible Party: Principal Investigator, Jeffrey Samet, Chief of General Internal Medicine, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H-33269; R01DA037768 (NIH)
Record Dates: First submitted 2015-09-28; First posted 2015-09-30 (Estimated); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: HIV Infection; Pain; Drug Dependence
Keywords: HIV Infection; Pain; Collaborative Care; Chronic Opioid Therapy; Addiction; Analgesics, Opioid
MeSH Terms: conditions — HIV Infections; Pain; Substance-Related Disorders; Behavior, Addictive | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TEACH Collaborative Care Intervention (Experimental): Physicians randomized to the intervention will receive: 1) collaboration with an IT enabled nurse care manager; 2) physician education and academic detailing; and 3) facilitated access to a specialist in addictions to help manage the most challenging HIV-infected patients on COT.
  Interventions: Behavioral: Collaboration with an IT enabled nurse care manager; Behavioral: Education and academic detailing; Behavioral: Facilitated access to a specialist in addictions
- Standard of Care Control (No Intervention): Physicians in the control group will receive information summarizing guidelines for COT but will not have access to the support of the TEACH intervention.

INTERVENTIONS:
Behavioral: Collaboration with an IT enabled nurse care manager — The nurse care manager at each site will collaborate with intervention physicians to implement key essential elements of guideline driven care, namely opioid treatment agreements, urine drug testing, random pill counts and periodic checking of on-line Prescription Monitoring Programs. The nurse care manager will use an electronic registry to retrieve pain medication information from the electronic medical record (EMR). Registry data will be collected on the patients of the intervention group providers. The nurse care manager will be able to use the registry to generate reports that will allow him/her to monitor those patients who are receiving opioids for chronic pain.
  Arms: TEACH Collaborative Care Intervention
Behavioral: Education and academic detailing — All intervention participants will receive a 60 minute group didactic session by a national expert on opioid prescribing for pain. Physicians will receive two academic detailing sessions, and will be given the option of having a third, booster academic detailing session if desired.
  Arms: TEACH Collaborative Care Intervention
Behavioral: Facilitated access to a specialist in addictions — The nurse care manager will encourage and arrange referral of challenging patients with potential abuse or dependence to prescription opioids to an addiction specialist.
  Arms: TEACH Collaborative Care Intervention

SUMMARY:
The TEACH randomized controlled trial will test the effectiveness of a collaborative care intervention directed towards physicians who provide care for HIV-infected persons to improve the quality of care for prescribing chronic opioid therapy (COT) for pain and reduce the misuse of prescription opioids among HIV-infected persons.

DETAILED DESCRIPTION:
The "Targeting Effective Analgesia in Clinics for HIV" (TEACH) Study will test the effectiveness of a collaborative care intervention directed toward HIV physicians to improve the management of chronic opioid therapy (COT) and reduce the misuse of prescription opioids among HIV-infected persons.

The intervention is composed of the following elements: 1) collaboration with an IT enabled nurse care manager; 2) physician education and academic detailing; and 3) facilitated access to a specialist in addictions to help manage the most challenging HIV-infected patients on COT. The nurse care manager will utilize an electronic registry to assist physicians in implementing guideline-driven care including opioid treatment agreements, urine drug testing (UDT), random pill counts and checking of online Prescription Monitoring Programs (PMPs). Physicians in the control group will receive information summarizing guidelines for COT but will not have access to the support of the TEACH intervention. This study is multi-site and will be conducted at Boston Medical Center and Grady Hospital (teaching hospital of Emory University). The 2-site study will use a cluster randomized trial design, randomized at the level of the physician, and compare primary outcomes over one year. The Specific Aims are to test the effectiveness of the TEACH collaborative care program to achieve the following: Aim 1 - to test whether the TEACH collaborative care program improves HIV physicians' adherence to guidelines for prescribing COT compared to standard practice; Aim 2 - to assess whether patient level outcomes improve as a result of the TEACH intervention; Aim 3 - to test whether the intervention increases HIV physicians' satisfaction with prescribing COT; and Aim 4 - to assess whether the intervention improves virologic control among HIV-infected patients who are on COT. If effective, implementation of the intervention in HIV clinics will enable physicians in clinical teams to deliver chronic opioid therapy according to established guidelines with more confidence, potentially resulting in less prescription drug abuse and improved HIV outcomes.

There are two distinct components to the study. The intervention, outlined in this Clinical Trials Protocol Registration and Results System (PRS) summary, involves consenting physicians as participants in a randomized controlled trial of an intervention and, via a waiver of informed consent, extracting patient level data on the physicians' patients from the electronic medical record. The patient cohort component, which is outlined in a separate Clinical Trials PRS summary, will involve recruiting and consenting patients in the HIV clinic on COT to be participants in an observational study, which will involve interviewing them to collect self-reported data and conducting medical chart reviews.

If effective, implementation of the TEACH intervention in clinics will enable physicians who provide primary care to HIV-infected patients in clinical teams to deliver chronic opioid therapy according to established guidelines with more confidence, potentially resulting in less prescription drug abuse and improved HIV outcomes.

ELIGIBILITY:
Physician Inclusion Criteria:

* Physician (i.e. MD, DO) or Advanced Practice Provider (i.e., Nurse Practitioner or Physicians Assistant) at enrollment sites.
* Main provider for ≥ 1 HIV-infected patient on COT (defined as having received ≥ 3 opioid prescriptions at least 21 days apart within a 6 month period).

Physician Exclusion Criteria:

* Investigator on this study.
* Planning to leave clinic < 9 months from enrollment.

Patient Inclusion Criteria:

* COT patient ages ≥ 18 who are patients of physicians enrolled in the TEACH study.

Patient Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Patient receipt of ≥2 UDT (Electronic Medical Record (EMR) extraction) | 12 Months
% of patients who have ≥1 early refill (i.e., any early refills) (EMR extraction) | 12 Months
Physician satisfaction managing HIV-infected patients on COT for pain (Physician self-report) | 12 Months

SECONDARY OUTCOMES:
≥3 primary care visits in infectious disease clinic (EMR extraction) | 12 Months
% of patients who had a discontinuation of their narcotic prescriptions (EMR extraction) | 12 Months
Opioid treatment agreement (EMR extraction) | 12 Months
% of physicians who self-report consulting the state Prescription Monitoring Program (Physician self-report) | 12 Months
Number (continuous measure) of early refills at 12 months (EMR extraction) | 12 Months
Patient aberrant use (Patient self-report) | 12 Months
Number of patients who have visited the emergency department to seek opioids (EMR extraction and patient self-report) | 12 Months
Patient pain severity and interference (Patient self-report) | 12 Months
Patient addiction severity (Patient self-report) | 12 Months
Physician confidence in prescribing COT (Physician self-report) | 12 Months
Patient satisfaction with COT (Patient self-report) | 12 Months
Patient trust in physician (Patient self-report) | 12 Months

OTHER OUTCOMES:
Undetectable HIV viral load (EMR extraction) | 12 Months
Cluster of differentiation 4 (CD4) cell count (EMR extraction) | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Samet, MD, MA, MPH, Principal Investigator — Boston Medical Center; Carlos del Rio, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University, Atlanta, Georgia
  - Boston Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ngo B, Liebschutz JM, Cheng DM, Colasanti JA, Merlin JS, Armstrong WS, Forman LS, Lira MC, Samet JH, Del Rio C, Tsui JI. Hazardous alcohol use is associated with greater pain interference and prescription opioid misuse among persons living with HIV and chronic pain. BMC Public Health. 2021 Mar 22;21(1):564. doi: 10.1186/s12889-021-10566-6. PMID 33752634
- [Derived] Lira MC, Tsui JI, Liebschutz JM, Colasanti J, Root C, Cheng DM, Walley AY, Sullivan M, Shanahan C, O'Connor K, Abrams C, Forman LS, Chaisson C, Bridden C, Podolsky MC, Outlaw K, Harris CE, Armstrong WS, Del Rio C, Samet JH. Study protocol for the targeting effective analgesia in clinics for HIV (TEACH) study - a cluster randomized controlled trial and parallel cohort to increase guideline concordant care for long-term opioid therapy among people living with HIV. HIV Res Clin Pract. 2019 Apr;20(2):48-63. doi: 10.1080/15284336.2019.1627509. PMID 31303143